CLINICAL TRIAL: NCT03809676
Title: Periodontal Status and Dental Behavior of Heart Trasplant Recipients and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yasemin Sezgin, asistant professor, Baskent University
Other Study IDs: BaskentU4
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Periodontal Diseases; Heart Transplantation
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- heaart transplant recipients
  Interventions: Other: periodontal examination
- healthy controls
  Interventions: Other: periodontal examination

INTERVENTIONS:
Other: periodontal examination — clinical measurements were recorded

SUMMARY:
Forty heart transplant recipients and forty age and sex mathced systemically healthy patients were included. Periodontal examination was performed and a questionnaire was applied to record demographic data, systemic health and dental behavior data.

DETAILED DESCRIPTION:
Patients who had heart transplantion surgery at between 2003 to 2017 were screened during routine outpatient visits. The patients who have history of periodontal treatment within the previous year, history of antibiotic use during the preceding 6 months, clinically non-stable patients were excluded . 40 cardiac transplant patiets who met these criteria included into this study. Each member of the transplant group was mathched with a patient in the systemically healthy control group by age and gender and smoking status. 40 systemically healthy subjects with no history of periodontal treatment within the previous year and no history of antibiotic use during the preceding 6 months were recruited.

Medical Data Hospital records were reviewed and data were collected using a standardised form that included demographic information (age, gender) and medical information such as smoking history, presence of systemic disease, post transplant time, medication regimen/dosages. Assesment of Oral Hygeine Behaviour Patients were also asked to complete a standardised anamnestic questionnaire. Questions were about their personal oral hygeine behaviour (toothbrush, dental floss etc.), whether their dental visit was routine or complaint-oriented. For the transplant group one more question about whether a dental check up or comprehensive dental treatment had occured before transplantation was added.

Clinical Examination In both groups, periodontal examination was performed by one calibrated periodontist at the Deperatment of Periodontology, Başkent University. All subjects recieved a comprehensive periodontal examination including plaque index (PI); gingival index (GI); gingival recession (GR); bleeding on probing (BOP); Probing depth (PD); clinical attachment level (CAL).

According to the clinical and radiographic evaluation the patients were categorized due to their periodontal status. The patients were diagnosed with periodontally healthy, gingivitis or periodontitis. Patients were diagnosed with periodontally healthy if they have <10% bleeding sites with probing depths ≤3 mm; whereas patients who have >10% bleeding sites with probing depths ≤3 mm were diagnosed with gingivitis. Patients who had probing depths ≥ 4 mm, interproximal, CAL of ≥2 mm or ≥3 mm at ≥2 non-adjacent teeth .9,25,26

ELIGIBILITY:
For transplant group:

Inclusion criteria:

* Having heart transplantation surgery
* be clinically stable

Exclusion criteria

* History of periodontal treatment within the previous year,
* history of antibiotic use during the preceding 6 months,
* being clinically non-stable For healthy group Inclusion criteria
* being systemically healthy
* no history of periodontal treatment within the previous year
* no history of antibiotic use during the preceding 6 months exclusion criteria Having a systemic disease

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: 40 transplant recipients and 40 systemically healthy patients were recruited
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
probing depth | day 1
  measured form pocket depth to the gingival margin by periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin Sezgin, Ankara, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No